CLINICAL TRIAL: NCT04708743
Title: The Tongue Features Associated With Chronic Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University, Taiwan (Other)
Responsible Party: Principal Investigator, Jia-Ming Chen, Principal Investigator, China Medical University, Taiwan
Other Study IDs: CCH
Record Dates: First submitted 2021-01-11; First posted 2021-01-14 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: CKD
Keywords: ATDS,Tongue Features

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CKD group: patients with CKD stage 3-5 including dialysis, followed tongue images by Automatic Tongue Diagnosis System
  Interventions: Diagnostic Test: Automatic Tongue Diagnosis System
- Health group: patients who had no past history or systemic disease, CKD followed tongue images by Automatic Tongue Diagnosis System
  Interventions: Diagnostic Test: Automatic Tongue Diagnosis System

INTERVENTIONS:
Diagnostic Test: Automatic Tongue Diagnosis System — tongue image capture tongue images by Automatic Tongue Diagnosis System

SUMMARY:
The Automatic Tongue Diagnosis System (ATDS) was developed to capture tongue images and extract features reliably to assist the diagnosis of TCM practitioners.This project will employ the ATDS verified to extract the tongue features of patients with chronic kidney disease(CKD) including dialysis patients. A TCM indices derived through the non-intrusive tongue diagnosis procedure can provide valuable information for clinical doctors to analyze the current status of a patient and dynamically schedule a treatment plan, facilitating early detection and diagnosis of CKD.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is an important global public health problem. According to related literatures, the prevalence of CKD is about 11% .CKD is a progressive disease. If it progresses to end-stage renal disease (ESRD), renal replacement therapy: dialysis and renal transplantation, is required to maintain life. The growing prevalence and progression of chronic kidney disease (CKD) raises concerns about our capacity to manage its economic burden to patients, caregivers, and society. The societal direct and indirect costs of CKD and end-stage renal disease are substantial and increase throughout disease progression. There is significant variability in the evidence about direct and indirect costs attributable to CKD and end-stage renal disease, with the most complete evidence concentrated on direct health care costs of patients with advanced to end-stage CKD.

CKD, also called chronic kidney failure, is described as a sustained reduction in glomerular filtration rate or evidence of structural or functional kidney abnormalities.Chronic kidney disease (CKD) refers to all five stages of kidney damage, from very mild damage in stage 1 to complete kidney failure in stage 5. CKD symptoms include pain, itch(pruritus), peripheral numbness, sleep disturbances, depression, fatigue, nausea and vomiting. Factors that contribute to these symptoms include anaemia, uraemic toxins, reduced renal capacity, chronic disease-related inflammation, and psychological stress associated with long-term illness.If it progresses to end-stage renal disease (ESRD), renal replacement therapy, including hemodialysis, peritoneal dialysis and kidney transplantation, is required to maintain life. Therefore, it is essential to find effective and conservative treatment methods to delay the progression of CKD.

Diagnosis in traditional Chinese medicine (TCM) is based on four procedures, observation, smelling or listening, inquiry, and palpation. Tongue diagnosis, serving as a vital non-invasive tool to provide useful clinical information, plays a pivotal role in TCM. The tongue is considered to reflect the physiological and pathological condition of the body, as well as the degree and progression of disease, through the meridians that connect the tongue to the internal organs.By observing tongue features, TCM practitioners can probe qi-blood, yin-yang disorders which are important in treatment selection and prognosis.Clinically, practitioners observe tongue characteristics, such as tongue color and shape, fur color and thickness, and the amount of saliva, to help deduce the primary pattern of a patient. However, tongue diagnosis is often biased by subjective judgment, which originates from personal experience, knowledge, diagnostic skills, thinking patterns, and color perception/interpretation.The inconsistency of subjective diagnosis can be improved by using the development of validated instruments. The automatic tongue diagnosis system (ATDS) has shown high consistency and can provide objective and reliable information and analysis of tongue features, facilitating doctors in making effective observations and diagnoses of specific diseases.Previous studies have been conducted on exploring the association between tongue characteristics and specific diseases, including rheumatoid arthritis, breastcancer,type 2 diabetes, metabolic syndrome, eczema, dysmenorrhea and functional dyspepsia, gastroesophageal reflux disease.However, to the best of our knowledge, no study has yet been performed on the comprehensive scrutiny of tongue features in patients with CKD using ATDS.

The objectives of this protocol are to apply the noninvasive ATDS to evaluate tongue manifestations in patients with CKD, and to provide valuable information for clinical doctors, which can be used to facilitate the early detection and diagnosis of CKD, to analyze the current status of patients, and to dynamically schedule treatment plans.

ELIGIBILITY:
Inclusion Criteria:

* age over 20 years old;
* CKD group:CKD stage 3-5 including dialysis patients
* Healthy group: without any medical history

Exclusion Criteria:

* cancer;
* acute infection;
* unable to protrude the tongue stably;
* risk of temporomandibular joint dislocation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with CKD stage3-5
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-05-19 (Actual); Primary Completion 2021-01-30 (Estimated); Study Completion 2021-04-20 (Estimated)

PRIMARY OUTCOMES:
Tongue features | 5 mins
  capture tongue images by Automatic Tongue Diagnosis System(ATDS)

CONTACTS AND LOCATIONS:
Overall Officials: Lun-Chien Lo, phd, Principal Investigator — School of Chinese Medicine, China Medical University, Taichung, Taiwan.
Locations (1):
- School of Chinese Medicine, China Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lo LC, Cheng TL, Chiang JY, Damdinsuren N. Breast cancer index: a perspective on tongue diagnosis in traditional chinese medicine. J Tradit Complement Med. 2013 Jul;3(3):194-203. doi: 10.4103/2225-4110.114901. PMID 24716178
- [Result] Lo LC, Chiang JY, Cheng TL, Shieh PS. Visual agreement analyses of traditional chinese medicine: a multiple-dimensional scaling approach. Evid Based Complement Alternat Med. 2012;2012:516473. doi: 10.1155/2012/516473. Epub 2012 Sep 17. PMID 23024693
- [Result] Lee TC, Lo LC, Wu FC. Traditional Chinese Medicine for Metabolic Syndrome via TCM Pattern Differentiation: Tongue Diagnosis for Predictor. Evid Based Complement Alternat Med. 2016;2016:1971295. doi: 10.1155/2016/1971295. Epub 2016 May 25. PMID 27313640
- [Result] Lo LC, Chen CY, Chiang JY, Cheng TL, Lin HJ, Chang HH. Tongue diagnosis of traditional Chinese medicine for rheumatoid arthritis. Afr J Tradit Complement Altern Med. 2013 Aug 12;10(5):360-9. doi: 10.4314/ajtcam.v10i5.24. eCollection 2013. PMID 24311851
- [Result] Lo LC, Chen YF, Chen WJ, Cheng TL, Chiang JY. The Study on the Agreement between Automatic Tongue Diagnosis System and Traditional Chinese Medicine Practitioners. Evid Based Complement Alternat Med. 2012;2012:505063. doi: 10.1155/2012/505063. Epub 2012 Aug 8. PMID 22924055
- [Result] Kim J, Son J, Jang S, Nam DH, Han G, Yeo I, Ko SJ, Park JW, Ryu B, Kim J. Availability of tongue diagnosis system for assessing tongue coating thickness in patients with functional dyspepsia. Evid Based Complement Alternat Med. 2013;2013:348272. doi: 10.1155/2013/348272. Epub 2013 Sep 15. PMID 24159343
- [Derived] Chen JM, Chiu PF, Wu FM, Hsu PC, Deng LJ, Chang CC, Chiang JY, Lo LC. The tongue features associated with chronic kidney disease. Medicine (Baltimore). 2021 Mar 5;100(9):e25037. doi: 10.1097/MD.0000000000025037. PMID 33655979

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-25): https://cdn.clinicaltrials.gov/large-docs/43/NCT04708743/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/43/NCT04708743/ICF_001.pdf